CLINICAL TRIAL: NCT03321331
Title: Can Commercial Mobile Apps for Weight Management be Used in Interventions? Bridging the Gap Between Usability, Theoretical Adherence, and User Experience - Part II - WaznApp Trial
Brief Title: A Self-directed Mobile Intervention to Promote Weight Control Among Employees of a Lebanese University
Acronym: WaznApp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Marco Bardus, Assistant Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: URB103369
Record Dates: First submitted 2017-10-11; First posted 2017-10-25 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Body Weight Changes; Overweight and Obesity; Sedentary Lifestyle; Health Behavior
Keywords: Mobile Health; mobile apps; weight control; weight management; self-directed intervention; behavioral intervention
MeSH Terms: conditions — Body Weight Changes; Overweight; Obesity; Sedentary Behavior; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessments regarding body weight and waist circumference will be conducted by nurses at the University Health Services clinics, who are blind to treatment allocation. The assessor will go through an assessment training program and will be informed about the study, but not about the allocation or treatments. Due to the nature of the intervention neither participants nor staff can be blinded to allocation, but are strongly inculcated not to disclose the allocation status of the participant at the follow up assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lark (JITAI) (Experimental): Participants in the intervention arm will use for 12 weeks the pro version of a mHealth app called "Lark", developed by Lark Technologies Ltd. Lark is a coach app, which uses several variables to generate smart and empathic conversations. Variables include activity, sleep, meals, weight, and height data, weight goal set by the user/Lark coach, activity goal set by user/Lark coach, starchy food goal set by user/Lark coach. Lark uses all these variables to create a dynamic coaching system, constantly changing and adapting to the user in the moment and over time. For these features, Lark provides a just in time adaptive intervention (JITAI).
  Interventions: Combination Product: Lark (JITAI)
- MyFitnessPal (no JITAI) (Active Comparator): Participants in the control arm will be assigned to use MyFitnessPal. Similar to the intervention arm, they will be instructed to use the app for 12 weeks. MyFitnessPal does not include JITAI components, but allows users to keep track of their caloric intake and energy expenditure. MyFitnessPal has features that can be associated with effective behavior change techniques, including: self-monitoring of behavior and outcomes, goal setting and feedback (similar to Lark). In MyFitnessPal, social support is limited to comments and 'likes' from friends of its restricted user community, therefore tackling the techniques of "social comparisons" and "social reward".
  Interventions: Combination Product: MyFitnessPal (no JITAI)

INTERVENTIONS:
Combination Product: Lark (JITAI) — Lark works as a just-in-time adaptive intervention (JITAI), providing interactive counseling through a chat-style interface. The app prompts users to self-monitor, set goals, review them, provides feedback, and social support.
  Other Names: Lark
  Arms: Lark (JITAI)
Combination Product: MyFitnessPal (no JITAI) — MyFitnessPal (MFP) is a calorie counting app, which relies on user input for food tracking, but automatically tracks activity through the phone or through integrations with wearable devices. This app provides allows to set weight and caloric goals, review them and to receive feedback, but it has limited social support, a feature that is generally lacking in calorie-counting apps.
  Other Names: MyFitnessPal
  Arms: MyFitnessPal (no JITAI)

SUMMARY:
WaznApp study is a 12-week randomized controlled trial aimed to evaluate the feasibility and preliminary efficacy of a self-directed behavioral weight-loss intervention targeting employees of an academic institution, using two popular consumer mobile applications for weight loss. The hypothesis is that individuals assigned to the app that provides interactive feedback and proactively motivates engagement in healthy behaviors (eating healthily and being more active) will be significantly better than those who receive the comparison condition (a simple calorie tracking app).

DETAILED DESCRIPTION:
BACKGROUND: Recent reviews show that popular mobile apps for weight loss and weight management embed elements that are commonly associated with behavior change, such as setting goals, self-reporting and monitoring behavior, and prompting feedback on performance. These technologies show good potential for developing interventions for the prevention of noncommunicable diseases. Despite their potential, little is known about how these changes can occur and the way end-users perceive and use these apps. Few studies tested if commercial apps for weight management can be used in interventions for behavior change.

PURPOSE: To assess the feasibility and preliminary efficacy of a self-directed weight-loss intervention targeting employees of an academic institution, using consumer mobile applications for weight loss (Lark and MyFitnessPal).

SETTING: American University of Beirut campus and Medical Center, Beirut, Lebanon.

PARTICIPANTS: Employees (adults aged 18+), with criteria of being able to read, write, and understand English, being owners of a mobile phone with either Android (v4.4 or above) or iPhone operative system (v8 or later); in better controlling their weight, and provide written informed consent to participate in the trial.

RESEARCH DESIGN: The study is a single-center, parallel randomized controlled trial with two study arms (intervention and control). The intervention arm will use Lark, a mobile coach app, which provides a just-in-time adaptive intervention (JITAI) by providing motivational feedback, goal setting, and emotional social support, among other change techniques. The control group will use MyFitnessPal, a calorie-counting app, which does not include JITAI components, but allows users to keep track of their caloric intake and energy expenditure.

EXPECTED IMPACT: This project will provide preliminary evidence on the efficacy of weight management apps, promoting behavior change among employees of an academic workplace. The results will inform larger scale studies targeting this population in Lebanon, and will be used as benchmark for further investigations in other settings and with other target groups.

ELIGIBILITY:
Inclusion Criteria:

1. Be an employee of the American University of Beirut (AUB) or its Medical Center (AUBMC).
2. To be able to read, write, and understand English.
3. To own a mobile phone with either Android (v4.4 or above) with or iOS (v8 or later).
4. To be interested in better controlling their weight.

Exclusion Criteria:

1. Students, who cannot prove their status as full-time or part-time employees at AUB or AUBMC.
2. Employees who are not able to read, write, and understand English.
3. Employees who do not own a mobile phone with either Android (v4.4 or above) or iOS (v8 or later).
4. Employees who have physical disabilities preventing them from exercising or walking.
5. Employees who are on a special diet for treatment of chronic conditions (e.g., Diabetes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Weight change (kg) | Baseline, 4, 8, 12 weeks
  Absolute change in weight (kg)
Waist circumference change (cm) | Baseline, 12 weeks
  Absolute change in waist circumference (cm)
BMI change (kg/m^2) | Baseline, 4, 8, 12 weeks
  Absolute change in BMI (kg/m^2)
Physical activity change (self-reported - IPAQ-SF, MET-hours/week) | Baseline, 12 weeks
  Measured through the International Physical Activity Questionnaire, short form (IPAQ-SF). IPAQ-SF requires respondents to estimate how much time they spent while doing activities in the previous week, in four domains: vigorous or moderate physical activity, walking and sitting. A total physical activity score is calculated by summing the time spent in each domain. Total physical activity score and sub-domain scores can be expressed in hours/week, or converted to metabolic-equivalents (METs), following the IPAQ scoring protocol.
Physical activity change (automatically tracked - steps/week) | Baseline, 4, 8, 12 weeks
  Through mobile phone accelerometer.
Dietary caloric intake change | Baseline, 12 weeks
  Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool, version 2016, developed by the National Cancer Institute, Bethesda, MD. The multiple pass approach in 24-hour recall consists of 8 modules: a meal based quick list, meal gap review, detail pass, final review, forgotten foods, last chance, usual intake question and supplements module. It provides a detailed assessment of dietary intake over the past 24 hours including food, drinks and supplements, as well as timing, form, portion size, the way food has been prepared, consumption of additions such as sugar, cream, dressing, etc., in addition to the source/brand of food. The 2016 version of the system includes also pictures of portions which are deemed to reduce overestimation or underestimation of food intake.

SECONDARY OUTCOMES:
Adherence | 4, 8, 12 weeks
  Number of missing data within each of the surveys.
Rate of Recruitment and Retention | 4, 8, 12 weeks
  Number of participants who were recruited, enrolled, successfully completed the study, and/or dropped out.
Program acceptability | 4, 8, 12 weeks
  Qualitative acceptability feedback related to the program will be collected at each data point through open-ended questions ("Do you have any concerns about the study procedures? Write a comment in the field below"; "Do you have any concerns about the app you have used? Write a comment in the field below"; "Do you have any concerns about the questionnaires? Write a comment in the field below")
Satisfaction with the program | 12 weeks
  7-point rating scale (semantic differential) ranging from extremely satisfied to extremely dissatisfied. An open-ended question will give participants the option to elaborate on their response.
Perceived app quality change (uMARS scale) | 4, 12 weeks
  App quality will be assessed through the user version of the Mobile App Rating Scale - uMARS. The uMARS scale provides a measure of app quality based on the average of four sub-domains: engagement, functionality, aesthetics, and information. Each of the sub-domains is based on the average value of multiple items, assessed through 5-point Likert scales (engagement: 5 items; functionality and information: 4 items; aesthetics: 3 items). The uMARS includes also 4 items that are aimed to address a subjective quality domain, which are: Would you recommend this app to people who might benefit from it? How many times do you think you would use this app in the future if it was relevant to you? Would you pay for this app? What is your overall star rating of the app?
Motivation to lose weight change (S-weight scale) | Baseline, 12 weeks
  Stages of change (S-Weight) scale.
Motivation to lose weight change (P-weight scales) | Baseline, 12 weeks
  Processes of change (P-Weight) scale.
Treatment Self-Regulation Questionnaire change (TSRQ scale) | Baseline, 4, 8, 12 weeks
  TSRQ measures the motivation to participate in the program. The TSRQ scale includes autonomous and controlled regulation subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bardus, PhD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- AUB Health & Wellness Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Bardus M, Hamadeh G, Hayek B, Al Kherfan R. A Self-Directed Mobile Intervention (WaznApp) to Promote Weight Control Among Employees at a Lebanese University: Protocol for a Feasibility Pilot Randomized Controlled Trial. JMIR Res Protoc. 2018 May 16;7(5):e133. doi: 10.2196/resprot.9793. PMID 29769174

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT03321331/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT03321331/ICF_001.pdf